CLINICAL TRIAL: NCT04274881
Title: Evaluation of Surface Landmarks and C-length as Predictors of the Depth of Right Internal Jugular Venous Catheter Insertion: A Transesophageal Echocardiography-Guided Study
Brief Title: Surface Landmarks and C-length as Predictors of Depth of Right IJV Catheter Insertion: A TEE-Guided Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh M. Hakim, Professor of Anesthesiology, Intensive Care and Pain Management, Ain Shams University
Other Study IDs: FMASU MS 301/2019
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Catheterization, Central Venous; Echocardiography, Transesophageal; Anatomic Landmarks; Radiography
Keywords: Surface landmarks; C-length; Central venous catheterization; Internal jugular vein; Prediction; Accuracy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheterization of internal jugular vein — The right internal jugular vein will be cannulated under transesophageal echocardiographic (TEE) guidance in order to place the catheter tip in the mid-SVC.
  The length of the catheter required to place the tip at the mid-SVC as guided by TEE will be regressed on the C-length or on the distance from the entry point to the surface point corresponding to the mid-SVC on the chest wall in order to obtain a predictive equation.
  The accuracy of either equation will be assessed by estimation of the standard error of the estimate (SEest).
  Other Names: Transesophageal echocardiography (to guide placement of central venous catheter tip at mid-SVC)

SUMMARY:
The primary aim of this study is to derive a prediction rule to estimate the required length for placement of the CVC tip at the mid-point of the SVC from simple anatomical landmarks that are consistent with the known surface projections of the great veins. The accuracy of this rule will be examined using TEE and is intended for adult patients undergoing cannulation of the right IJV utilizing a middle approach. As a secondary aim, we will examine the performance of this suggested rule as contrasted with two other popular methods for estimation of the CVC length, the Peres formula and the C-length method.

DETAILED DESCRIPTION:
Before induction of anesthesia

Three sets of measurements will be obtained for each participant before induction of anesthesia:

1. Surface measurements: Three points will be placed on the skin using a non-erasable marker. Point A, at the apex of the triangle between the two heads of the sternomastoid. Point B, at the ipsilateral sternoclavicular joint. Point C, at the lower border of the right 2nd rib at its junction with the sternum. The distance between point A and point B and between point B and point C will be measured and added to each other to determine the catheter length expected to place the tip at the mid-SVC.
2. Radiological measurements: On the plain posteroanterior (PA) chest X-ray (CXR), the distance from the tip of the transverse process of T1 to the tracheal bifurcation (C-length) will be measured.
3. Using Peres' formuls (Height in cm/10), we will record the anti After induction of anesthesia After induction of anaesthesia, the TEE probe will be placed and a bicaval view will be displayed to visualize the right atrium-superior vena cava (RA-SVC) junction and the proximal (lower) part of the SVC at its entry into the right atrium (RA). The TEE probe will be manipulated to display the SVC as far as possible from its junction with the RA.

The right internal jugular vein (IJV) will be cannulated under ultrasound guidance using the Seldinger technique.

After puncture of the IJV a J-wire will be advanced through the trocar until the J-end of the guidewire is visualized at the RA-IJV junction via the TEE.

The CVC catheter will be passed over the guidewire to the RA-SCV junction. The guidewire will be removed and the catheter will then be retracted under TEE guidance until the tip in visualized at 3.0 cm above the RA-SVC junction as measured with the TEE cursor. If the distal (upper) portion of the SVC could not be visualized, the catheter would be retracted for 3 cm as guided by the 1-cm gradations on the CVC.

Post-operative After operation, plain PA CXR will be obtained at the intensive care unit (ICU) to verify the position of the CVC tip in relation to the carina.

Statistical Analysis:

The length of the catheter required to place the tip at the mid SVC will be regressed on the C-length or the surface distance to obtain a predictive equation. The accuracy of either equation will be assessed by estimation of the standard error of the estimate (SEest).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (age 18 years or older).
* Elective cardiac surgery.
* Echocardiography is indicated or recommended.

Exclusion Criteria:

* Previous cardiothoracic or neck surgery.
* Previous radiotherapy on the neck or chest.
* Intra-thoracic or neck mass lesions.
* Deformity of the chest wall.
* Anomalies of the great vessels.
* Congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects of either sex who are scheduled for elective cardiac surgery in whom echocardiography is indicated or recommended will be eligible.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of surface landmarks for prediction of CVC depth required to place the CVC tip at the mid-SVC. | Outcome will be assessed at completion of catheterization procedure
  Difference between actual length required to place the CVC tip at the mid-SVC as guided by TEE and the distance from the entry point to the surface point corresponding to the mid-SVC on the chest wall.
Accuracy of C-length for prediction of CVC depth required to place the CVC tip at the mid-SVC. | Outcome will be assessed at completion of catheterization procedure
  Difference between actual length required to place the CVC tip at the mid-SVC as guided by TEE and the C-length.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M Hakim, MD, Study Director — Ain Shamd University, Faculty of Medicine, Department of Anesthesiology
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No